CLINICAL TRIAL: NCT00142246
Title: Intermittent Preventive Treatment in Schools: a Randomised Controlled Trial of the Impact of IPT on Malaria, Anaemia and Education Amongst Schoolchildren in Western Kenya
Brief Title: Study of the Impact of Intermittent Preventive Treatment in Schools on Malaria, Anaemia and Education.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITDCVG41
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Malaria, Falciparum
Keywords: malaria; anaemia; school performance; education; intermittent preventive treatment; schools
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Anemia | interventions — Amodiaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intermittent preventive treatment with antimalarial drug combination(SP and amodiaquine)
  Interventions: Drug: Intermittent preventive treatment (SP and amodiaquine)
- 2 (Placebo Comparator): Dual placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intermittent preventive treatment (SP and amodiaquine) — Oral medication. SP: single dose given over one day; amodiaquine: 3 daily doses over 3 days. Dosage has given according to age.
  Arms: 1
Other: Placebo — Three doses given over three days (Day 1: placebo SP + placebo AQ; Days 2 and 3: placebo AQ). Dosage given according to age
  Arms: 2

SUMMARY:
This study seeks to establish whether intermittent preventive treatment (IPT) can reduce malaria among school-going children and its consequent impact on school performance.

DETAILED DESCRIPTION:
Although the risk of malaria is greatest in early childhood, significant numbers of schoolchildren remain at risk from malaria-specific morbidity and mortality. Each year between 20-50% of schoolchildren, aged 10-14 years, living in malaria-endemic areas will experience a clinical attack of malaria (Clarke et al., 2004). Malaria accounts for 3-8% of all-cause absenteeism from school, and up to 50% of preventable absenteeism (Brooker et al., 2000). In addition, asymptomatic parasitaemia contributes to anaemia, reducing concentration and learning in the classroom (Holding & Snow, 2001). Intermittent preventive treatment (IPT) delivered through schools is a simple intervention, which can be readily integrated into broader school health programmes. This study seeks to examine whether IPT can reduce malaria and anaemia amongst school-going children, and its consequent impact on school performance, in order to assess its suitability for inclusion as a standard intervention in school health programmes.

The efficacy of IPT is being evaluated in schoolchildren with a high-level of acquired immunity and ability to limit parasite growth, in whom most infections are asymptomatic and may go untreated.

The intervention: Intermittent preventive treatment of malaria administered each school term with the purpose to reduce asymptomatic parasitaemia and prevent clinical attacks, thereby reducing anaemia and school absenteeism, with consequences for improved attendance and concentration in class.

Schools are randomly allocated to one of two arms:

* Intervention schools: IPT given three times a year (once per term) + mass treatment with anthelminthics
* Control schools: mass treatment with anthelminthics only

Mass treatment with anthelminthics is carried out in all study schools twice annually in accordance with national policy.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in primary school, and attending regularly
* Enrolled in nursery or classes 1-7
* Informed consent from parent or guardian

Exclusion Criteria:

* Enrolled in primary class 8
* Haemoglobin level below 70g/L at baseline
* History of reaction to sulfa drugs (e.g. fansidar, septrin)
* History of severe skin reaction to any drug

Withdrawal criteria:

* Withdrawal of parental consent
* Haemoglobin level falling below 70g/L
* Severe adverse reaction to treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6758 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of anaemia (Hb <112g/L) | March 2006

SECONDARY OUTCOMES:
Prevalence of Plasmodium falciparum parasitaemia | March 2006
Sustained attention | March 2006
Mean haemoglobin | March 2006

CONTACTS AND LOCATIONS:
Overall Officials: Sian E Clarke, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine, University of London, UK; Simon J Brooker, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine, University of London, UK; Benson BA Estambale, MBChB, PhD, Principal Investigator — University of Nairobi; Matthew CH Jukes, PhD, Principal Investigator — Partnership for Child Development, Imperial College, University of London, UK; Pascal Magnussen, MD, Principal Investigator — DBL - Institute for Health Research and Development, Denmark
Locations (1):
- Primary schools within Bondo district / Bondo District Hospital, Bondo, Bondo District, Kenya

REFERENCES:
- [Background] Clarke SE, Brooker S, Jukes MCH, Njagi JK, Khasakhala L, Otido J, Crudder C, McGlone B, Magnussen P & Estambale BBA. (2006). Randomised controlled trial of intermittent preventive treatment in schoolchildren: Impact on malaria, anaemia & school performance [abstract]. American Journal of Tropical Medicine & Hygiene Suppl 75 (5): 123.
- [Background] Clarke S, Njagi J, Jukes M, Estambale B, Khasakhala L, Ajanga A, Luoba A, Otido J, Ochola S & Magnussen P. (2005). Intermittent preventive treatment in schools: Malaria parasitaemia, anaemia and school performance [abstract]. Acta Tropica, Suppl 95: S133.
- [Derived] Clarke SE, Jukes MC, Njagi JK, Khasakhala L, Cundill B, Otido J, Crudder C, Estambale BB, Brooker S. Effect of intermittent preventive treatment of malaria on health and education in schoolchildren: a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2008 Jul 12;372(9633):127-138. doi: 10.1016/S0140-6736(08)61034-X. PMID 18620950